CLINICAL TRIAL: NCT03155230
Title: Nationwide Results on Chronic Pain After Bilateral Transabdominal Preperitoneal Inguinal Hernia Repair (TAPP)
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Niels Johansen, Principal Investigator, Hvidovre University Hospital
Other Study IDs: nj01042017
Record Dates: First submitted 2017-05-14; First posted 2017-05-16 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Hernia, Inguinal; Chronic Pain
Keywords: Inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Danish male patients who had undergone bilateral TAPP (July 2012 to June 2013) were recruited from the Danish Hernia Database and cross-checked with hospital files and the National Patient Registry. A standardized postal questionnaire was sent out two years after the index surgery to investigate Patients Related Outcome Measures (PROMs) such as chronic post-operative pain.

DETAILED DESCRIPTION:
The present study was primarily undertaken to provide evidence for the risk of activity-related chronic postoperative inguinal pain following bilateral TAPP in an all-male Danish setting. Impaired sexual activity and sleep disturbance due to pain was also recorded. Data based on nationwide consecutive patients undergoing bilateral TAPP. Data collected for the Danish Inguinal Hernia Database, hospital files and the National Patient Registry (Denmark).

ELIGIBILITY:
Inclusion Criteria:

* Danish males,
* Age>18 years
* Elective, bilateral TAPP due to inguinal hernia within the period from July 1, 2012 to June 30 2013

Exclusion Criteria:

* age <18 years
* miss-classified surgical code
* non-Danish speaking
* psychiatric anamneses
* regarded and non-compliant patients who had either died, emigrated or were lost to follow-up emergency repair
* femoral hernia repair

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Danish males, age>18 years undergoing elective, bilateral TAPP due to inguinal hernia (medial, lateral, and combined hernias) within the study period from July 1, 2012 to June 30 2013
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Activities Assessment Scale Questionnaire | Within one week
  Impaired daily activities by chronic pain from either one or both groin areas

SECONDARY OUTCOMES:
Questionnaire about sexual impairment | Within three months
  Sexual impairment due to chronic pain from either one or both groin areas
Questionnaire about sleep impairment | Within three months
  Sleep impairment due to chronic pain from either one or both groin areas

CONTACTS AND LOCATIONS:
Overall Officials: Thue Bisgaard, professor, Study Director — HvidovreUT
Locations (1):
- Gastrounit, Surgical Division, Hvidovre Hospital, Denmark, Copenhagen, Danmark, Denmark